CLINICAL TRIAL: NCT00432107
Title: A Multi-centre, Two-stage, Open Label Phase II Study to Assess the Efficacy and Safety of APO866 in the Treatment of Patients With Advanced Melanoma.
Brief Title: A Study to Assess APO866 for the Treatment of Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP3003
Record Dates: First submitted 2007-02-06; First posted 2007-02-07 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2013-11

CONDITIONS: Melanoma
Keywords: Advanced cutaneous melanoma; Phase II study
MeSH Terms: conditions — Melanoma | interventions — N-(4-(1-benzoylpiperidin-4-yl)butyl)-3-(pyridin-3-yl)acrylamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2-stage mono therapy of APO866 (Experimental): The treatment period consists of 3 consecutive 28 day cycles. Each cycle starts with a 4 day continuous infusion of the study medication followed by a 24 day break
  Interventions: Drug: APO866

INTERVENTIONS:
Drug: APO866 — APO866 is administered as 0.126 mg/m²/hr IV every 4 weeks for 4 consecutive days (96 hours) for a total of 3 cycles

SUMMARY:
This phase II study is designed to determine the efficacy and safety of APO866 for the treatment of patients with advanced cutaneous melanoma. APO866 has shown to induce growth inhibition in cultures of human melanoma cells as well as in animal models with subcutaneously implanted melanoma tumors. APO866 was considered to be safe and well tolerated in a phase I study that treated 24 patients with advanced cancer. In that study one of the two patients with advanced melanoma had a stable disease for 5 months with size reduction of some lesions. APO866 is administered by intravenous infusion continuously for 96 hours that is repeated every 4 weeks. Patients will receive 3 cycles of treatment and the primary efficacy endpoint will be assessed at Week 16. Patients will be follow-up for 12 months.

DETAILED DESCRIPTION:
Advanced melanoma is one of the most chemo-resistant types of human cancers. The incidence increases by about 2.5% on an annual basis, with may partially be related to aging and growth of the population, as well as other environmental risk factors. Virtually no recent progress has been made in the treatment of patients with this disease. In the past 30 years, the FDA has approved only 2 agents, dacarbazine and interleukin-2, on the basis of overall response and response duration, respectively. However, these outcomes were not accompanied by a survival benefit. The most recent randomized study of Dacarbazine (DTIC) yielded an overall response rate of 7%, and to date, no other treatments, including combination therapies, have shown to improve survival when compared to DTIC alone. Hence, the mainstay of treatment for patients with advanced melanoma is DTIC-based therapy.

APO866 is a novel drug that induces cell death by specifically inhibiting the biosynthesis of Niacinamide Adenine Dinucleotide (NAD+) from niacinamide, which is essential for the cellular metabolism, protein modification and messenger synthesis. APO866 is not subject to the commonly known mechanisms of multi drug resistance (MDR). Its activity is cell cycle independent. APO866 exerted high anti-tumor activity on a broad range of different tumor cells derived from both human solid cancers and leukemias in vitro and on a large number of human xenografts in nude mice, including melanoma, and rats in vivo. Hematologic cancer cells were highly sensitive to APO866. Lymphocytes are the most sensitive normal cells to APO866 resulting in lymphocytopenia and reticulocytopenia in rats, monkeys. Furthermore, APO866 may have anti-angiogenic properties as shown in vivo.

APO866 was investigated in 24 patients with advanced cancers in a phase I study aiming to determine the dose-limiting toxicity (DLT) and maximum tolerated dose (MTD). Treatment was well tolerated and safe. The unique DLT was thrombocytopenia. At dose levels higher than 0.036 mg/m2/hr CTC grade III lymphocytopenia, not thought to be clinically relevant, preceded all other toxicities. The recommended dose for phase II studies of APO866 is 0.126 mg/m2/hr administered by civ infusion for 4 consecutive days evry 4 weeks. This dose was selected because of its safety profile, and the translational observation that Css of APO866 at MTD was similar or higher as compared to the concentrations at which efficacy was established in vitro and in vivo. In addition, a transient decrease of serum vascular endothelial growth factor (VEGF) levels, a surrogate marker of angiogenesis, was observed within 96 hrs after the start of treatment in 9 out of 11 patients treated at MTD and the 0.144 mg/m2/hr dose level of APO866.

No objective tumor response was observed. However, 4 patients had stable disease for at least 3 months: prostate cancer (4 months), melanoma (5 months), sarcomatoid mesothelioma (3 months) and oropharyngeal cancer (5 months). In addition, lesion size reductions were observed in the melanoma patient (80% size reduction and stable size of other lesions) at an APO866 dose level of 0.072 mg/m2/hr, and in the mesothelioma patient (moderate size reductions of pleural lesions) at 0.108 mg/m2/hr.

Treatment with APO866 was safe and well tolerated. The anti-tumor effect of APO866, in particular on melanoma cells in vitro and in vivo, and its anti-angiogenic propriety support the rationale to conduct a open phase II study of APO866 in patients with advanced melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of melanoma
* Stage IV disease or stage III not amenable to surgery (AJCC, see Appendix A)
* Measurable disease, defined as at least 1 malignant lesion that could be accurately and serially measured in at least 1 dimension and for which the greatest diameter is > or = 10 mm as measured by spiral computed tomography (CT) scan or magnetic resonance imaging (MRI), or > or = 20 mm with conventional techniques. A caliper can be used for the measurement of superficial cutaneous metastases which are > or = 10 mm.
* Patients must be able to undergo either contrast-enhanced CT-scan or contrast-enhanced MRI scan for tumor assessment
* Only one previous systemic treatment (excluding prior systemic treatment as postoperative adjuvant therapy) is allowed and should have been terminated > 4 weeks before Study Day 1 (SD1).
* Lack of response or progression of disease after the most recent systemic therapy for advanced melanoma
* Patients must have recovered from the toxicity of any previously used treatment. All Adverse events of previous systemic treatment must have resolved to < grade I Common Terminology Criteria for Adverse Events (CTC v3.0, see Appendix)
* Eastern Cooperative Oncology Group (ECOG) Performance Status < 1 (see Appendix C)
* Age > 18 years, of either sex
* Female patients with childbearing potential must be using a hormonal contraceptive, intra uterine device, diaphragm with spermicide or condom with spermicide for the duration of the study. Women of childbearing potential must have a negative serum or urinary human chorionic gonadotropin (hCG) pregnancy test within 7 days prior to Study Day 1 (SD1)
* Male patients, who are not surgically sterile, must use a condom with spermicide for the duration of the study and 3 months thereafter
* Have given written informed consent, prior to any study related procedure not part of the patient's normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

* Have participated in any other investigational study or received an experimental therapeutic procedure considered to interfere with the study in the 4 weeks preceding SD1
* History of brain metastases or leptomeningeal disease
* Bone-only metastatic disease
* Use of prohibited medication due to Cytochrome P450 3A4 (CYP3A4) metabolism of APO866, as specified in Section 6.6.2. concomitant use of these drugs will not be allowed during the study.
* Use of biphosphonate drug during the 30 days preceding the APO866 infusion and during the treatment period will not be allowed
* Uncontrolled medical conditions, requiring surgical or pharmacological treatment (exceptions must be approved by the Medical Responsible of the study).
* Serious concomitant disease (e.g. significant cardiac disease)
* History of second cancer that was treated with curative intent and in complete remission for < 5 years, with the exception of basal cell carcinoma or cervical cancer in situ
* Primary or acquired thrombocytopenia
* Inadequate bone marrow reserve: white blood cell (WBC) < 3.5x10^9/L, neutrophils < 1.0x10^9/L, thrombocytes < 100x10^9/L, Hb < 10.0 g/dL or coagulation abnormalities
* Inadequate liver function: total bilirubin > 1.5 x upper limit of normal values (ULN), aspartate aminotransferase (AST), Alanine Amino Transferase (ALT), or alkaline phosphatase > 2.5 x ULN
* Have inadequate renal function, defined by serum creatinine > 1.5x ULN
* Retinopathy, history of retinal laser surgery, or an ERG < 50% of normal
* Pregnant of lactating female
* Abuse of alcohol or other recreational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-07; Primary Completion 2008-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To determine the tumor response rate (according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria) as the proportion of eligible patients with stage IV cutaneous melanoma or stage III not amenable to surgery. | Week 16

SECONDARY OUTCOMES:
Safety and tolerability | Week 16 and 12 months follow-up
Time to response | Week 16
Duration of response | Week 16
Progression free survival | 12 months
Overall survival | 12 months
Evolution of serum VEGF and interleukin-8 (IL-8) during treatment | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Trefzer, MD PhD, Principal Investigator — Department of Dermatology, Charité University Hospital, Schumannstrasse 20-21, 10117 Berlin, Germany
Locations (6):
- Department of Dermatology, Medical University Graz, Graz, Austria
- France (2):
  - Department of Dermatology, Hopital Henri Modor, Créteil
  - Department of Dermatologie, Hotel Dieu, Nantes
- Germany (2):
  - Department of Dermatology, Charité University Hospital Berlin, Berlin
  - University Clinic for Dermatology, Medical Faculty of Mannheim of the Heidelberg University, Mannheim
- Department of Dermatology, University Hospital of Zürich, Zurich, Switzerland